CLINICAL TRIAL: NCT06976905
Title: Myoma Screw in Manipulation of Large Uterus in Total Laparoscopic Hysterectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mona Gamil, Resident, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KFSIRB200-545
Record Dates: First submitted 2025-04-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Total Laparoscopic Hysterectomy With Myoma Screw

STUDY DESIGN:
Intervention Model Description: 1 group using uterine manipulator vs another group using myoma screw
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myoma screw usage in total laparoscopic hysterectomy in large uterus (Experimental): Using myoma screw from abdominal approach in manipulation Instead of traditional uterine mani Pulator
  Interventions: Procedure: Total laparoscopic hysterectomy
- Uterine manipulator in total laparoscopic hysterectomy in large uterus (Experimental): Using traditional uterine manipulator via vagina in uterine manipulation
  Interventions: Procedure: Total laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Total laparoscopic hysterectomy — Hysterectomy by laparoscope using uterine manipulator or myoma screw as a manipulator of large uterus

SUMMARY:
To compare between myoma screw and uterine manipulator in manipulation of large uterus in total laparoscopic hysterectomy

DETAILED DESCRIPTION:
Hysterectomy is performed on 1,500,000 women worldwide each year to treat benign disorders such leiomyoma, prolapse, and irregular bleeding, as well as gynecologic malignancies. Prior to the introduction of the first laparoscopic procedures in the late 1980s, hysterectomy was traditionally accomplished by laparotomy or the vaginal route. Total laparoscopic hysterectomy (TLH) became the most commonly used hysterectomy technique in the last ten years, especially in developed nations, because laparoscopic hysterectomy has some advantages over other hysterectomy types, including high patient satisfaction, an earlier return to work, less blood loss, the ability to diagnose and treat other pelvic diseases, and the ability to maintain thorough intraperitoneal haemostasis.

However, there are some drawbacks to TLH as well, such as its expensive cost, lengthier operating time, and requirement for advanced technological instruments including uterine manipulators (UM) and sealing devices.

In order to facilitate colpotomy by defining the cervicovaginal junction and enable safer dissection around the cervix, the main goal of utilising a UM is to extend the distance between the cervix and ureter.There isn't enough clinical data in the literature to say whether using UM meets these expectations, though.Additionally, the use of UMs has been linked to a number of specific problems, such as uterine rupture, intestinal perforation, and vaginal wall laceration.UMs are also not appropriate in certain cases, such as vaginal stenosis, anatomical differences that make it difficult to identify the uterus or cervix, and patients who refuse vaginal penetration because they are virgins. There is still no "optimal UM" that is consistently safe, effective, and economical, despite the fact that numerous UMs have been developed in recent decades.

Some studies have suggested alternatives including the use of certain sutures, gripping forceps, or myoma screws (MS) as answers to the issues that arise with the use of UM. When performing a myomectomy using the vaginal method, laparotomy, or laparoscopy, the MS is a conventional, reusable instrument. MSs are renowned for their ability to deliver a powerful three-dimensional traction force. Additionally, using MS does not require specialised knowledge like UMs do.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-60
2. BMI 25-40
3. Large uterus with fundal level 12-24w diagnosed by TAS( Transabdominal Ultrasound)/TVUS(Transvaginal ultrasound)
4. Adenomyosis

Exclusion Criteria:

1. BMI more than 40
2. patients with contraindication for laparscopic surgery e.g cardiac and cirrhotic patients

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Comparison between Magneshkar uterine manipulator and myoma screw in operation time in hours | During surgery in hours
  Using myoma screw as a manipulator in total laparoscopic hysterectomy

SECONDARY OUTCOMES:
Volume of blood loss in ml liters | Day 1
  Volume of blood loss in ml liters

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Egypt